CLINICAL TRIAL: NCT04041804
Title: Activation Intervals Effects on Non-surgical Semi-rapid Maxillary Expansion in Adults
Brief Title: Activation Intervals Effects on Non-surgical Maxillary Expansion in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Sonia Patricia Plaza, Director, Research Orthodontic Department, Principal Investigator., Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 044
Record Dates: First submitted 2019-02-13; First posted 2019-08-01 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Maxillary Anomaly
Keywords: Palatal Expansion Technique; Cone-Beam Computed Tomography
MeSH Terms: interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Every week RPE activation (Active Comparator): Non-surgical semi-rapid maxillary expansion (SRME) with the time intervals activation every week until getting the require expansion needed
  Interventions: Procedure: semirapid maxillary expansion (SRME)
- Every four days RPE activation (Active Comparator): Non-surgical semi-rapid maxillary expansion (SRME) with the time intervals activation every four days until getting the require expansion needed
  Interventions: Procedure: semirapid maxillary expansion (SRME)

INTERVENTIONS:
Procedure: semirapid maxillary expansion (SRME) — A Banded Hyrax is going to be used in order to provide an increase in the maxillary transverse dimension
  Other Names: Maxillary Expansion

SUMMARY:
OBJECTIVE: To evaluate the effects of different time intervals activations on the non-surgical maxillary expansion in adults. Methods: This study will include two groups, 10 adult patients each (mean age 20-35) with maxillary transverse deficiency and unilateral or bilateral crossbite. In the first group, the expansion is going to be activated every four days. In the second group, activation will occur every eight days. The primary outcomes are transverse dimension, the buccal cortical bone formation, and the upper premolar and molar labial inclination. Dentoalveolar changes will be evaluated using CBCT images and digital models.

ELIGIBILITY:
Inclusion Criteria

* Presence of transverse maxillary deficiency unilateral or bilateral in which the maxillary cusps of at least two premolars and/or maxillary molars occluded on the central fossa of the antagonist's teeth
* The needs of maxillary expansion for the correction of their malocclusion
* Age range from 20 to 35
* Non-gingivitis or untreated caries at the start of orthodontic treatment
* Probing depth less than 4mm across the entire dentition
* Gingival index ≤ 1
* Plaque index ≤ 1

Exclusion Criteria:

* Increased Monson curve
* Patients with systemic disease
* Patients with congenital anomalies
* Medicated patients (long term use of antibiotics, Phenytoin, cyclosporine, anti-inflammatory drugs, systemic corticosteroids, and calcium channel blockers)
* Pregnancy
* Poor oral hygiene for more than two visits
* Radiographic evidence of moderate to severe bone loss
* Current periodontal disease
* Patients who smoke
* Individuals with inadequately treated endodontic problems in the study area.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Transversal distance between upper canines, first premolars and upper first molars | Change from baseline to 6 months
  Distance between mesial fosa of each upper canines, first premolars and distance between central fosa of each upper first molars
Posterior teeth buccal inclination | Change from baseline to 6 months
  Measure in CBCT in a coronal slice between the palatal plane and the dental axis
Buccal bone area evaluation | Change from baseline to 6 months
  Measure in CBCT in a coronal slice, thickness of the buccal bone in upper first premolars and upper first molars

SECONDARY OUTCOMES:
Bleeding on probing (BP) | Change from baseline to 6 months
  It's going to be measured by clinical exam with a periodontal probe and it is verified the presence of bleeding and it will be register as 0= No bleeding and 1= bleeding
Evaluation of the perception of pain by the patient (VAS) | Change from baseline to 6 months
  Pain visual analogue scale (AVS) - from 0 to 10 points, Higher values represent more pain perception by the participant
Probing depth (PD) | Change from baseline to 6 months
  Probing depth (PD): It's going to be measured by clinical exam with a periodontal probe and it is measured from the gingival margin to the bottom of the groove. It is considered the presence of a periodontal pocket when the depth of the groove is greater than 3mm.
Clinical attachment level (CAL) | Change from baseline to 6 months
  Linear measurement in mm. It is constructed from the relationship between probe depth (PD) and the measurement in millimeters from the cement enamel junction (CEJ) to the gingival margin
Soft tissue recession (STR) | Change from baseline to 6 months
  Soft tissue apical migration of the cement-enamel junction, it is going to classified as:
  Class I: Retraction of marginal tissue that does not extend to the mucogingival junction without loss of interdental tissue.
  Class II: Retraction of marginal tissue that extends to the mucogingival junction, or beyond it, there is no loss of bone, nor of interdental soft tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Arango, DDS, Study Chair — Fundación Universitaria UniCIEO
Locations (1):
- Fundación Universitaria UniCIEO, Bogotá, DC, Colombia